CLINICAL TRIAL: NCT02127073
Title: Identifying the miR Fingerprint in NAF, Serum, and Tissue in Patients With Ductal Carcinoma in Situ (DCIS) or Invasive Breast Cancer
Brief Title: Pilot Study of Oxytocin and microRNA Identification in NAF, Serum, and Tissue in Women With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Could not identify collaborator and secure additional funding after transferring the record to Montefiore Medical Center
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AAAL5203
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Results first posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Ductal Carcinoma in Situ
Keywords: Breast cancer; Ductal carcinoma in situ (DCIS); Oxytocin
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxytocin (Experimental): Subjects would receive 4 IU of intranasal oxytocin; one spray in each nostril, single-use.
  Interventions: Drug: Intranasal Oxytocin

INTERVENTIONS:
Drug: Intranasal Oxytocin — Intranasal spray, one spray or 4 IU of oxytocin will be administered into each nostril of each patient about 15-30 minutes before NAF collection
  Other Names: Syntocinon Spray

SUMMARY:
The purpose of this study is to examine the genetic material called microRNA of three types of specimens from women with breast cancer. The study also seeks to examine the effectiveness of using a new agent called oxytocin to increase the amount of nipple fluid that can be collected during surgery.

DETAILED DESCRIPTION:
Vast majority of breast cancers arise from ductal epithelium. Ductal cells can be collected through the nipple orifice very early in breast cancer development. The nipple aspirate ﬂuid (NAF) can be used to identify biomarkers that predict risk of breast cancer. To date, the biomarkers identified in nipple aspirate ﬂuid (NAF) have limited utility due to the large volume of NAF required for data analysis. Recent studies show intranasal oxytocin's utility in enhancing the yield of nipple aspirate ﬂuid (NAF) among healthy, non-lactating female patients as well as those at high risk for breast cancer. This capability is crucial for the analysis of various markers associated with breast disease and cancer such as microRNAs. The primary aim of the study is to determine whether the microRNA profile characterization is feasible with the collection of tissue, serum and NAF in patients with in situ and invasive breast cancer. Intranasal oxytocin will be used to enhance ﬂuid yielding of the NAF.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Ductal carcinoma in situ (DCIS) or invasive breast cancer
* Candidate for breast conserving surgery or mastectomy

Exclusion Criteria:

* Pregnant women
* Prior Breast Cancer diagnosis
* Adverse reaction to Oxytocin in the past

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-01-30 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Feldman, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial officially opened to enrollment in 2015 with first patient enrolled on 1/30/2015 at Columbia University Medical Center.
Period: Overall Study
Arm/Group | Oxytocin
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oxytocin
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Detection of microRNA in NAF, Serum, or Tissue
Time Frame: 3 years
Population: The study was voluntarily suspended as documented in IND Annual Report (Serial Number 0007). Data was not collected/aggregated and no interim analyses were conducted.
Arm/Group | Oxytocin
Number analyzed (Participants) | 0

2. Secondary Outcome: Percentage of Patients With Collection of ≥ 5 μL of Nipple Aspirate Fluid
Time Frame: 3 years
Population: as for outcome 1
Arm/Group | Oxytocin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From initiation of any study procedures to the end of the study treatment follow-up period at the Visit 2/End of Study visit, up to 4 weeks
Arm/Group | Oxytocin
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/73/NCT02127073/Prot_SAP_000.pdf